CLINICAL TRIAL: NCT02278380
Title: In-Vivo Glycemic Index (GI) and Insulinemic Index (II) Testing of 7 Test Foods in Total (5 Milk-based Beverage and 2 Standard Breakfast Items)
Brief Title: Different Glycemic Index (GI) Values in 7 Food Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: GDM.1.C/D
Record Dates: First submitted 2014-09-12; First posted 2014-10-30 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): To compare the Glycemic Index value of seven test foods:
  Low GI standard Breakfast Medium GI standard Breakfast Nutritional pregnant milk supplement Nutritional product for diabetics Pregnant and lactation women milk powder Nutritional drinks for diabetics Test product
  Interventions: Other: Low GI Standard Breakfast; Other: Medium GI Standard Breakfast; Other: Enfamama A+; Other: Glucerna Triple Care; Other: Dumex Precima; Other: Diasip; Other: Test product

INTERVENTIONS:
Other: Low GI Standard Breakfast — Low GI Standard Breakfast
Other: Medium GI Standard Breakfast — Medium GI Standard Breakfast
Other: Enfamama A+ — Nutritional pregnant milk supplement
Other: Glucerna Triple Care — Nutritional product for diabetics
Other: Dumex Precima — Pregnant and lactation women milk powder
Other: Diasip — Nutritional drinks for diabetics
Other: Test product — Test product not patented yet
  Other Names: Not patented yet, cannot disclose name.

SUMMARY:
This study is initiated to investigate the glycemic index value of seven food products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant females at least 6 weeks postpartum, non-lactating and aged 21-60yrs old in both groups.
* They should not suffer from any chronic diseases.
* no known food allergy or intolerance.
* no medications known to affect glucose tolerance(excluding oral contraceptives). Note: stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable.

Exclusion Criteria:

* Age less than 21 years old and greater than 60 years old.
* known history of diabetes mellitus or the use of antihyperglycemic drugs or insulin to treat diabetes and related conditions.
* known history of AIDS, hepatitis, renal or heart disease or any other serious complications that may interfere with glucose metabolism.
* subjects using any medication (eg steroids, protease inhibitors or antipsychotics, etc.) that would interfere with the digestion and nutrient absorption.,
* subjects having gastrointestinal diseases that may interfere with nutrient absorption, distribution, metabolism, excretion and have no known food allergies.
* a major medical or surgical event requiring hospitalisation within the preceding 3 months.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Glycemic index values of all seven products | 120 minutes post administration
  Glycemic index values at 120 minutes post adminstration.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Bhaskaran, Dr, Principal Investigator — Temasek Polytechnic
Locations (1):
- Temasek Polytechnic, Singapore, Singapore